CLINICAL TRIAL: NCT00599690
Title: Epi-LASIK : A Confocal Microscopy Analysis of the Corneal Epithelium and Anterior Stroma.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Asociación para Evitar la Ceguera en México, Asociación para Evitar la Ceguera en México
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Cornea 3
Record Dates: First submitted 2008-01-08; First posted 2008-01-24 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Corneal Epithelium
Keywords: Epi-LASIK-LASIK microkeratome; Corneal thickness; Confocal microscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Epithelial flaps were created with the Amadeus II, epi-LASIK-LASIK microkeratome (Ziemer ophthalmics systems AG, Switzerland). A Visx star 4 system (Visx, Santa Ana, CA, USA) was used to perform the laser ablation in all eyes
  Interventions: Procedure: Epi-LASK

INTERVENTIONS:
Procedure: Epi-LASK — 10 eyes of 10 patients underwent epi-LASK, epithelial flaps were created with the Amadeus II, epi-LASIK-LASIK microkeratome (Ziemer ophthalmics systems AG, Switzerland). A Visx star 4 system (Visx, Santa Ana, CA, USA) was used to perform the laser ablation in all eyes

SUMMARY:
To evaluate the confocal microscopy findings at the corneal epithelium and anterior stroma after epi-LASIK Surgery.

DETAILED DESCRIPTION:
10 eyes of 10 patients underwent epi-LASK, epithelial flaps were created with the Amadeus II, epi-LASIK-LASIK microkeratome (Ziemer ophthalmics systems AG, Switzerland). A Visx star 4 system (Visx, Santa Ana, CA, USA) was used to perform the laser ablation in all eyes. A central scan of the total corneal thickness was taken with the confocal microscope (Confoscan 4, Fortune Technologies, Italy) before and at 2 weeks and 1 month after surgery. Corneal epithelial thickness and the Anterior stroma morphology were analyzed by using the NAVIS software V. 3.5.0 (NIDEK, Multi-Instrument Diagnostic System, Japan).

ELIGIBILITY:
Inclusion Criteria:

* Patients asking for epi-LASIK surgery
* Patients with stable refraction in the last year
* Patients without systemic and ocular disease
* Patients with 500 microns in pachymetry
* Normal topography

Exclusion Criteria:

* Patients cannot attend their appointments
* Residual, recurrent or active ocular disease
* Previous ocular surgery except LASIK
* Autoimmune or connective tissue disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
A central scan of the total corneal thickness was taken with the confocal microscope (Confoscan 4, Fortune Technologies, Italy) | Before and at 2 weeks and 1 month after surgery

SECONDARY OUTCOMES:
There are no secondary outcome measures specified for this study | There are no secondary outcome measures specified for this study

CONTACTS AND LOCATIONS:
Overall Officials: Ramirez F Manuel, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación Para Evitar la Ceguera en Mëxico, Hospital "Luis Sánchez Bulnes"., Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Kollias A, Ulbig MW, Spitzlberger GM, Abdallat WH, Froehlich S, Welge-Luessen U, Lackerbauer CA. Epi-LASIK using the Amadeus II microkeratome: evaluation of cut quality using light and electron microscopy. J Cataract Refract Surg. 2007 Dec;33(12):2118-21. doi: 10.1016/j.jcrs.2007.07.038. PMID 18053914
- [Background] Gamaly TO, El Danasoury A, El Maghraby A. A prospective, randomized, contralateral eye comparison of epithelial laser in situ keratomileusis and photorefractive keratectomy in eyes prone to haze. J Refract Surg. 2007 Nov;23(9 Suppl):S1015-20. doi: 10.3928/1081-597X-20071102-07. PMID 18047000
- [Background] Katsanevaki VJ, Kalyvianaki MI, Kavroulaki DS, Pallikaris IG. One-year clinical results after epi-LASIK for myopia. Ophthalmology. 2007 Jun;114(6):1111-7. doi: 10.1016/j.ophtha.2006.08.052. Epub 2007 Feb 23. PMID 17320960
- [Background] Hoang-Xuan T, Arnaud D, Souissi K, Cornu S. [Epi-LASIK, a novel surface photoablation technique]. J Fr Ophtalmol. 2007 May;30(5):535-8. doi: 10.1016/s0181-5512(07)89639-2. French. PMID 17568349